CLINICAL TRIAL: NCT05354388
Title: Ripretinib Combined With Surgery in Advanced Gastrointestinal Stromal Tumors That Have Failed Imatinib Therapy: A Multicenter,Observational Study
Brief Title: Ripretinib Combined With Surgery in Advanced GIST That Have Failed Imatinib Therapy: A Multicenter,Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Minghui Pang, Professor, Sichuan Provincial People's Hospital
Other Study IDs: 20211013
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Gastrointestinal Stromal Tumor(GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgery after ripretinib treatment: For subjects who achieved PR or SD, perform resection of gastrointestinal stromal tumor
  Interventions: Procedure: Resection surgery of gastrointestinal stromal tumor

INTERVENTIONS:
Procedure: Resection surgery of gastrointestinal stromal tumor — oral administration of Ripretinib 150 mg QD. Resection of gastrointestinal stromal tumors was performed in patients who achieved PR or SD

SUMMARY:
The objective of this observational study is to explore the efficacy and safety of ripretinib treatment combined with surgery in advanced gastrointestinal stromal tumors(GIST) after failure of imatinib therapy.

DETAILED DESCRIPTION:
This study is a single-arm, multicenter, observational study. A total of approximately 30 subjects were be enrolled. The patient was orally administered with ripretinib150 mg QD. 4 weeks for one cycle. Efficacy was assessed every two cycles. For subjects with PR or SD after ripretinib treatment, resection of gastrointestinal stromal tumor was performed after discussion by MDT and ensure R0 resection as much as possible.Ripretinib 150mg QD was continued 2 weeks after surgery. Thereafter, subjectss entered the follow-up period for at least 1 year. Safety and survival information will be collected

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily, and signed a written informed consent, good compliance with follow-up;
2. 18 years ≤ age < 75 years, male or female;
3. Histopathological examination confirmed the diagnosis of recurrent and/or metastatic advanced unresectable gastrointestinal stromal tumor;
4. According to the modified RECISTv1.1-GIST-specific criteria, the subject has at least one measurable lesion;
5. Subjects must have progressed on imatinib or have documented intolerance to imatinib.
6. ECOG PS of ≤ 2, ASA score ≤ 3 at screening;
7. No other malignant tumors occurred within five years;

Exclusion Criteria:

1. Molecular pathology report PDGFRA Exon 18 mutation(including D842v);
2. Patients with other serious complications who cannot tolerate surgery: such as severe cardiopulmonary disease, heart function below clinical class 2, pulmonary infection, moderate to severe COPD, chronic bronchitis, severe diabetes and/or renal insufficiency, severe hepatitis and/or Child-pugh class C or B whose symptoms are significantly difficult to correct, severe malnutrition, etc;
3. Pregnant or lactating women;
4. Treatment with any other line of therapy in addition to imatinib for advanced GIST. Imatinib-containing combination therapy in the first-line treatment should not be enrolled.
5. Subject has known active central nervous system metastases.
6. Occurrence of bleeding, perforation, obstruction and other disease-related complications, requiring emergency surgery;
7. The patient has participated in or is participating in other clinical studies , or is taking other TKI agents;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled in this study will be outpatients from Sichuan Provincial People's Hospital and cooperative hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year Progression free survival rate | 12 monthes
  PFS Based on radiographic assessment using Choi criteria

SECONDARY OUTCOMES:
objective response rate（ORR） | 12 monthes
  Objective response rate as determined by confirmed CR + confirmed PR by radiologic review
R0 resection rate | 1 days after surgery
  R0 is the proportion of subjects with no microscopic residual after resection
2-year overall survival rate | 24 monthes
  Proportion of subjects with an overall survival time of at least 2 years
time to progression (TTP) | 12 monthes
  The time from the start of treatment to the progression
Duration of continuous medication before surgery | 12 monthes
  Only for subjects undergoing surgery

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Pang, Professor, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubin BP, Heinrich MC, Corless CL. Gastrointestinal stromal tumour. Lancet. 2007 May 19;369(9574):1731-41. doi: 10.1016/S0140-6736(07)60780-6. PMID 17512858
- [Background] Wozniak A, Rutkowski P, Piskorz A, Ciwoniuk M, Osuch C, Bylina E, Sygut J, Chosia M, Rys J, Urbanczyk K, Kruszewski W, Sowa P, Siedlecki J, Debiec-Rychter M, Limon J; Polish Clinical GIST Registry. Prognostic value of KIT/PDGFRA mutations in gastrointestinal stromal tumours (GIST): Polish Clinical GIST Registry experience. Ann Oncol. 2012 Feb;23(2):353-60. doi: 10.1093/annonc/mdr127. Epub 2011 Apr 28. PMID 21527588
- [Background] Reichardt P. The Story of Imatinib in GIST - a Journey through the Development of a Targeted Therapy. Oncol Res Treat. 2018;41(7-8):472-477. doi: 10.1159/000487511. Epub 2018 Jun 13. PMID 29895025
- [Background] Sciot R, Debiec-Rychter M, Daugaard S, Fisher C, Collin F, van Glabbeke M, Verweij J, Blay JY, Hogendoorn PC; EORTC Soft Tissue and Bone Sarcoma Group; Italian Sarcoma Group; Australasian Trials Group. Distribution and prognostic value of histopathologic data and immunohistochemical markers in gastrointestinal stromal tumours (GISTs): An analysis of the EORTC phase III trial of treatment of metastatic GISTs with imatinib mesylate. Eur J Cancer. 2008 Sep;44(13):1855-60. doi: 10.1016/j.ejca.2008.06.003. Epub 2008 Jul 22. PMID 18653326
- [Background] Bucher P, Villiger P, Egger JF, Buhler LH, Morel P. Management of gastrointestinal stromal tumors: from diagnosis to treatment. Swiss Med Wkly. 2004 Mar 20;134(11-12):145-53. doi: 10.4414/smw.2004.10530. PMID 15106018
- [Background] Martin-Broto J, Moura DS. New drugs in gastrointestinal stromal tumors. Curr Opin Oncol. 2020 Jul;32(4):314-320. doi: 10.1097/CCO.0000000000000642. PMID 32541319
- [Background] Dhillon S. Ripretinib: First Approval. Drugs. 2020 Jul;80(11):1133-1138. doi: 10.1007/s40265-020-01348-2. PMID 32578014
- [Background] Mantese G. Gastrointestinal stromal tumor: epidemiology, diagnosis, and treatment. Curr Opin Gastroenterol. 2019 Nov;35(6):555-559. doi: 10.1097/MOG.0000000000000584. PMID 31577561
- [Background] Serrano C, George S. Recent advances in the treatment of gastrointestinal stromal tumors. Ther Adv Med Oncol. 2014 May;6(3):115-27. doi: 10.1177/1758834014522491. PMID 24790651
- [Background] Bannon AE, Klug LR, Corless CL, Heinrich MC. Using molecular diagnostic testing to personalize the treatment of patients with gastrointestinal stromal tumors. Expert Rev Mol Diagn. 2017 May;17(5):445-457. doi: 10.1080/14737159.2017.1308826. Epub 2017 Mar 27. PMID 28317407
- [Background] Den Hollander D, Van der Graaf WTA, Desar IME, Le Cesne A. Predictive factors for toxicity and survival of second-line sunitinib in advanced gastrointestinal stromal tumours (GIST). Acta Oncol. 2019 Nov;58(11):1648-1654. doi: 10.1080/0284186X.2019.1637017. Epub 2019 Jul 26. PMID 31345082
- [Background] Janku F, Abdul Razak AR, Chi P, Heinrich MC, von Mehren M, Jones RL, Ganjoo K, Trent J, Gelderblom H, Somaiah N, Hu S, Rosen O, Su Y, Ruiz-Soto R, Gordon M, George S. Switch Control Inhibition of KIT and PDGFRA in Patients With Advanced Gastrointestinal Stromal Tumor: A Phase I Study of Ripretinib. J Clin Oncol. 2020 Oct 1;38(28):3294-3303. doi: 10.1200/JCO.20.00522. Epub 2020 Aug 17. PMID 32804590
- [Background] Blay JY, Serrano C, Heinrich MC, Zalcberg J, Bauer S, Gelderblom H, Schoffski P, Jones RL, Attia S, D'Amato G, Chi P, Reichardt P, Meade J, Shi K, Ruiz-Soto R, George S, von Mehren M. Ripretinib in patients with advanced gastrointestinal stromal tumours (INVICTUS): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Jul;21(7):923-934. doi: 10.1016/S1470-2045(20)30168-6. Epub 2020 Jun 5. PMID 32511981